CLINICAL TRIAL: NCT04247724
Title: The Physiological Health Effects of 12 Weeks of Small-sided Team Handball Training in Young Adult Women and Men
Brief Title: The Health Effects of Small-sided Team Handball
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Arne Astrup, Therese Hornstrup Bondebjerg, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H-15008361
Record Dates: First submitted 2020-01-20; First posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active group of men (Experimental): 4 groups are randomized for 12 weeks of intervention; 2 groups are active, 2 groups are inactive:
  *1 group of men playing recreational handball
  Interventions: Behavioral: Recreational handball
- Active group of women (Experimental): 4 groups are randomized for 12 weeks of intervention; 2 groups are active, 2 groups are inactive:
  *1 group of women playing recreational handball
  Interventions: Behavioral: Recreational handball
- Inactive group of men (Experimental): 4 groups are randomized for 12 weeks of intervention; 2 groups are active, 2 groups are inactive:
  *1 group of men continuing their normal lifestyle patterns
  Interventions: Behavioral: Control
- Inactive group of women (Experimental): 4 groups are randomized for 12 weeks of intervention; 2 groups are active, 2 groups are inactive:
  *1 group of women continuing their normal lifestyle patterns
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Recreational handball
  Arms: Active group of men; Active group of women
Behavioral: Control
  Arms: Inactive group of men; Inactive group of women

SUMMARY:
The purpose of the project was to examine the fitness and health effects of participation in recreational Team Handball for untrained 20-30 year old healthy men and women.

DETAILED DESCRIPTION:
Fitness and health effects of 12 weeks of recreational team handball in untrained adult men and women aged 20-30 years"

Adult men and women aged 20-30 years will be recruited to take part in a 12-week intervention with recreational team handball. Half of the participants are men (n=32), who are randomly assigned to a group playing recreational team handball (n=16) and an inactive control group (n=16). The women (n=40) are also divided and assigned to a group with regular participation in recreational team handball (n=20) and an inactive control group (n=20). The training sessions will be offered 2-3 times weekly for 70 minutes per session by a supervised trainer. The sessions involves an injury preventive warm-up and ball exercises for 15 minutes followed by recreational handball on small pitches such as 4 vs 4. A comprehensive testing protocol is conducted before and after the training period. The measurements includes body composition and bone mineralization, blood pressure, resting heart rate, fasting blood sugar, insulin, cholesterol and bone markers. In addition, a number of physical tests which involves fitness level (VO2max), intermittent work, muscle strength and balance will further be conducted. The testing takes place at the University of Copenhagen. The training sessions will also take place at the University of Copenhagen or in a handball club near the University. The study will be approved by the local ethical committee of Copenhagen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women and men from 20-30 years old
* If women, a regular menstrual cycle length (25 to 32 days) with or without use of contraceptives.

Exclusion Criteria:

* Known familiar diseases
* If been smoking for the last two years before recruitment
* If involved in any regular physical training two years before recruitment
* Women: a peak oxygen uptake (VO2peak) higher than 45 mL/min/kg
* Men: a peak oxygen uptake (VO2peak) higher than 51 mL/min/kg

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
VO2max - change is being assessed after 12 weeks of intervention | Measured before and after 12 weeks of intervention
  VO2max (mL/kg/min) is a measure of the cardiorespiratory during a treadmill test

SECONDARY OUTCOMES:
Fat percentage - change is being assessed after 12 weeks of intervention | Measured before and after 12 weeks of intervention
  Measure of fat percentage (%) performed by a dual energy x-ray absorptiometry (DXA scan)
Muscle mass - change is being assessed after 12 weeks of intervention | Measured before and after 12 weeks of intervention
  Measure of muscle mass (kg) performed by a DXA scan
Mineral bone density - change is being assessed after 12 weeks of intervention | Measured before and after 12 weeks of intervention
  Mineral bone density (g/cm2) performed by a DXA scan
Bone mass - change is being assessed after 12 weeks of intervention | Measured before and after 12 weeks of intervention
  Bone mass (kg) performed by a DXA scan

OTHER OUTCOMES:
Strength: Isokinetic Maximal voluntary contraction (MVC) - change is being assessed after 12 weeks of intervention | Measured before and after 12 weeks of intervention
  Isokinetic MVC (Nm) performed in a isokinetic dynamometer
Strength: Isometric MVC - change is being assessed after 12 weeks of intervention | Measured before and after 12 weeks of intervention
  Isometric MVC (Nm) performed in a isokinetic dynamometer
Strength: Countermovement maximal jumps (CMJ) jump height - change is being assessed after 12 weeks of intervention | Measured before and after 12 weeks of intervention
  CMJ jump height (cm) performed on a force plate
Strength: CMJ jump height - change is being assessed after 12 weeks of intervention | Measured before and after 12 weeks of intervention
  CMJ peak (W/kg) performed on a force plate
Postural balance: Sway area - change is being assessed after 12 weeks of intervention | Measured before and after 12 weeks of intervention
  Sway area (cm2) performed on a force plate
Postural balance: Sway length - change is being assessed after 12 weeks of intervention | Measured before and after 12 weeks of intervention
  Sway length (mm) performed on a force plate
Citrate synthase (CS) activity - change is being assessed after 12 weeks of intervention | Measured before and after 12 weeks of intervention
  Muscle biopsies were taken from the male subjects and analyzed for CS activity (ug/l)
3-hydroxyacyl-coenzyme A (CoA) dehydrogenase (HAD) activity - change is being assessed after 12 weeks of intervention | Measured before and after 12 weeks of intervention
  Muscle biopsies were taken from the male subjects and analyzed for HAD activity (ug/l)
Specific fibre type cross sectional area (CSA) - change is being assessed after 12 weeks of intervention | Measured before and after 12 weeks of intervention
  Muscle biopsies were taken from the male subjects and analyzed for specific fibre type CSA (μm2)
Fiber type composition - change is being assessed after 12 weeks of intervention | Measured before and after 12 weeks of intervention
  Muscle biopsies were taken from the male subjects and analyzed for fibre type composition (%)
Capillaries (cap./fiber) - change is being assessed after 12 weeks of intervention | Measured before and after 12 weeks of intervention
  Muscle biopsies were taken from the male subjects and analyzed for cap./fibre
Capillaries (cap./mm2) - change is being assessed after 12 weeks of intervention | Measured before and after 12 weeks of intervention
  Muscle biopsies were taken from the male subjects and analyzed for cap./mm2

REFERENCES:
- [Derived] Fristrup B, Krustrup P, Andersen JL, Hornstrup T, Lowenstein FT, Larsen MA, Helge JW, Povoas SCA, Aagaard P. Effects of small-sided recreational team handball training on mechanical muscle function, body composition and bone mineralization in untrained young adults-A randomized controlled trial. PLoS One. 2020 Nov 18;15(11):e0241359. doi: 10.1371/journal.pone.0241359. eCollection 2020. PMID 33206670